CLINICAL TRIAL: NCT04081376
Title: Generation of Biological Samples Positive to Hydromorphone for Anti-doping Control
Acronym: HM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IMIMFTCL/HM
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-09

CONDITIONS: Healthy Volunteers
Keywords: Hydromorphone; Opiates; Anti-doping control
MeSH Terms: interventions — Hydromorphone

STUDY DESIGN:
Intervention Model Description: There is one single treatment group (HM), and no control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Subjects receive a single-dose treatment.Urine samples will be collected after administration (8 fractions: 0-4h, 4-8h, 8-12h, 12-24h, 24-36h, 36-48h, 48-60h, 60-72h post-administration).
  Interventions: Drug: Hydromorphone Hydrochloride

INTERVENTIONS:
Drug: Hydromorphone Hydrochloride — 4 mg of hydromorphone hydrochloride (equivalent to 3.56 mg of hydromorphone) administered orally in a single dose.

SUMMARY:
Background:

Hydromorphone (HM) is a semi-synthetic derivative of morphine used for pain control. Like other opiates, due to its high potential of abuse HM is included on the World Anti-Doping Agency (WADA) list of prohibited substances.

Hypothesis:

The oral administration of hydromorphone hydrochloride in healthy subjects allows generating detectable concentrations of the drug in urine. Positive urine samples will enable to identify analytical strategies for doping control.

Objectives:

Primary objective: To measure the concentrations of hydromorphone in urine for anti-doping control samples.

Secondary objective: To identify metabolites and precursors of hydromorphone in urine. To assess safety and tolerability of the drug used.

Methods:

Phase I, open, non-randomized clinical trial, with a treatment condition (hydromorphone) administered orally to 2 subjects.

DETAILED DESCRIPTION:
This study aims to characterize the patterns of urinary excretion of HM following the oral administration of 4 mg of hydromorphone hydrochloride (equivalent to 3.56 mg of hydromorphone). The detection of HM consumption can be done by urine immunoassay but several immunoassay tests are required to thoroughly detect synthetic, semi-synthetic and natural opioids due to the limited cross-reactivity of each assay. Therefore, superior test strategies are required to specifically identify low concentrations of opioids.

ELIGIBILITY:
Inclusion Criteria:

* Male volunteers aged between 18 and 45 years.
* Able to understand and accept the trial procedures and able to sign an informed consent.
* History and physical examination that demonstrate not presenting organic or psychiatric disorders.
* ECG, blood and urine tests performed before the test within normal limits. Minor or occasional variations of these limits will be allowed if, in the opinion of the Principal Investigator and taking into account the state of science, they have no clinical significance, do not pose a risk to the subject and do not interfere in the product evaluation. These variations and their non-relevance will be specifically justified sin writing.
* Body mass index (weight/height^2) between 19 and 25 kg/m2. BMI between 25 and 27 kg/m2 may be included according to Principal Investigator's criteria.

Exclusion Criteria:

* History of allergy, idiosyncrasy, hypersensitivity or adverse reactions to the active substance or similar nonapeptides, or to any of the excipients.
* Patients who have undergone surgical interventions and/or have had underlying diseases that could lead to a stricture of the gastrointestinal tract, that have "blind handles" of the gastrointestinal tract or gastrointestinal obstruction.
* Patients with severe decrease in liver function.
* Patients with respiratory failure or history of asthma crisis.
* Patients with acute abdominal pain of unknown origin.
* Background or clinical evidence of gastrointestinal, hepatic, renal disorder or others that may involve an alteration of the absorption, distribution, metabolism or excretion of the drug, or that are suggestive of gastrointestinal irritation by drugs.
* Background or clinical evidence of psychiatric disorders, alcoholism, drug abuse or habitual consumption of psychoactive drugs.
* Having participated in another clinical trial with medication in the three months prior to the start of the study.
* Having suffered some organic disease or major surgery in the six months prior to the start of the study.
* Antecedents or clinical evidence of cardiovascular, respiratory, renal, hepatic, endocrine, gastrointestinal, hematological, neurological or other acute or chronic diseases that, in the opinion of the Principal Investigator or the collaborators designated by him/her, may pose a risk to the subjects or may interfere with the objectives of the study. Especially epileptic seizures or a history of epilepsy.
* Having taken medication regularly in the month prior to the study sessions. Treatment with monoamine oxidase inhibitors (MAOIs), buprenorphine, nalbuphine or pentazocine during the two months prior to the study. Treatment with single doses of another type of symptomatic medication in the week prior to the study sessions will not be a reason for exclusion if it is assumed that the drug has been completely eliminated on the day of the experimental session.
* Smokers of more than 20 cigarettes a day in the 3 months before the study.
* Consumption of more than 20 g of alcohol daily in women and more than 40 g in men.
* Consumers of more than 5 coffees, teas, cola drinks, or other stimulant drinks or with xanthines daily in the 3 months prior to the study start.
* Being unable to understand the nature, consequences of the trial and the procedures that are asked to follow.
* Positive serology for hepatitis B, C or HIV.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-18 (Actual)

PRIMARY OUTCOMES:
Urine concentration of hydromorphone | 0-4 hours post-administration
  Concentration of hydromorphone in fraction-1 urine samples
Urine concentration of hydromorphone | 4-8 hours post-administration
  Concentration of hydromorphone in fraction-2 urine samples
Urine concentration of hydromorphone | 8-12 hours post-administration
  Concentration of hydromorphone in fraction-3 urine samples
Urine concentration of hydromorphone | 12-24 hours post-administration
  Concentration of hydromorphone in fraction-4 urine samples
Urine concentration of hydromorphone | 24-36 hours post-administration
  Concentration of hydromorphone in fraction-5 urine samples
Urine concentration of hydromorphone | 36-48 hours post-administration
  Concentration of hydromorphone in fraction-6 urine samples
Urine concentration of hydromorphone | 48-60 hours post-administration
  Concentration of hydromorphone in fraction-7 urine samples
Urine concentration of hydromorphone | 60-72 hours post-administration
  Concentration of hydromorphone in fraction-8 urine samples

SECONDARY OUTCOMES:
Urine concentration of hydromorphone metabolites | 0-4 hours post-administration
  Concentration of different hydromorphone metabolites in fraction-1 urine samples
Urine concentration of hydromorphone metabolites | 4-8 hours post-administration
  Concentration of different hydromorphone metabolites in fraction-2 urine samples
Urine concentration of hydromorphone metabolites | 8-12 hours post-administration
  Concentration of different hydromorphone metabolites in fraction-3 urine samples
Urine concentration of hydromorphone metabolites | 12-24 hours post-administration
  Concentration of different hydromorphone metabolites in fraction-4 urine samples
Urine concentration of hydromorphone metabolites | 24-36 hours post-administration
  Concentration of different hydromorphone metabolites in fraction-5 urine samples
Urine concentration of hydromorphone metabolites | 36-48 hours post-administration
  Concentration of different hydromorphone metabolites in fraction-6 urine samples
Urine concentration of hydromorphone metabolites | 48-60 hours post-administration
  Concentration of different hydromorphone metabolites in fraction-7 urine samples
Urine concentration of hydromorphone metabolites | 60-72 hours post-administration
  Concentration of different hydromorphone metabolites in fraction-8 urine samples

CONTACTS AND LOCATIONS:
Overall Officials: Ana M Aldea Perona, Dr, Principal Investigator — IMIM (Hospital del Mar Medical Research Institute)
Locations (1):
- IMIM (Hospital del Mar Medical Research Institute), Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No